CLINICAL TRIAL: NCT02049463
Title: Advanced Analysis of the Carotid Phonoangiography and Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Chairman, National Taiwan University Hospital
Other Study IDs: 201311042RIND
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Carotid Atherosclerosis; Seeing Sounds as Colors; Stenosis; Stroke
Keywords: carotid artery; sound; stenosis; wall; stroke
MeSH Terms: conditions — Carotid Artery Diseases; Constriction, Pathologic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To investigate the different sound spectrum of carotid arteries and to analyze its relationship to the vessel disease, and to build a new biomarker about vascular disorder.

Methods: To record the carotid phonoangiography with digital stereoscopy and analysis the spectrum with different algorithm such as FFT, wavelet, entropy, complexity, and HHT. The results will be correlated and comparison to the finding in clinical, carotid Doppler and duplex, CTA, MR, and catheter angiography.

Statistics:

The significance of difference between parameters was computed using t-tests or paired t-test etc. A p value <0.05 is defined as significant.

DETAILED DESCRIPTION:
The investigators plan to recruit data from patients that come to their department for angiography study and intervention (n=300) with different disease entity such as atherosclerosis, tumor, aneurysm, arteriovenous malformation or fistula, and other vascular disorders. A period of about 20 seconds of the carotid phonoangiography was recorded.

Standard for comparison: catheter angiography, CTA, MRI/MRA. The degree of stenosis, the wall thickness, SI and density change was clustered and compared. The clinical and laboratory data will be reviewed and the vascular risk factors will be calculated.

Spectrum analysis: The sound spectrum will be analysis with the FFT, wavelet, entropy, complexity, and HHT algorithms.

The correlation between change of spectrums and also the correlated clinical, images, and laboratory change will be further analysis by statistic method.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 years old to 99 years old
2. Gender: Unlimited
3. Because different types of brain diseases, those who received conventional catheter vascular examination.

Exclusion Criteria:

1. Neck inflammation locally who can not admit the sound.
2. Due to inability to cooperate to accept those recordings.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who is going to have carotid angiography study and with informed consent signed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
progression of stenosis | three years
  Follow-up the severity of the carotid stenosis and correlate its wall change

SECONDARY OUTCOMES:
wall change | three years
  correlate the phonographic change with the follow up CTA wall change.

CONTACTS AND LOCATIONS:
Overall Officials: Hon-man Liu, MD, MBA, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Hon-Man Liu, Dawan, Taiwan, Taiwan